CLINICAL TRIAL: NCT03136159
Title: The Role of Adherent Occlusive Antimicrobial Absorbent Foam Dressing in Prevention of Cesarean Section Wound Complications
Brief Title: The Role of Antimicrobial Foam Dressing in Prevention of Cesarean Section Wound Complications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loyola University (Other)
Collaborators: Molnlycke Health Care AB (Industry)
Responsible Party: Principal Investigator, Jean Goodman, Director of Maternal Fetal Medicine, Loyola University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 207526
Record Dates: First submitted 2017-04-27; First posted 2017-05-02 (Actual); Results first posted 2020-12-21 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Cesarean Section; Complications, Wound, Dehiscence
Keywords: pregnancy; delivery; cesarean section; wound healing; silver-containing dressing
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Silver-impregnated antimicrobial dressing (Experimental): All participants undergoing primary cesarean section will receive a silver impregnated antimicrobial wound dressing (Mepilex Border AG), postoperative.
  Interventions: Device: Silver-impregnated antimicrobial dressing

INTERVENTIONS:
Device: Silver-impregnated antimicrobial dressing — All participants will receive an adherent soft silicone silver impregnated anti-microbial occlusive foam dressing after cesarean section. The dressing will stay on for up to seven days.
  Other Names: Mepilex Border AG

SUMMARY:
Post-cesarean section wound infections are responsible for longer hospital stays, readmissions, and ultimately, increased costs to the healthcare system. Silver-containing dressings may prevent wound infections. The purpose of the current study is to determine if the use of a silver-impregnated dressing decreases the occurence of wound infection following cesarean delivery.

DETAILED DESCRIPTION:
A single-centered, single-arm clinical trial was originally designed to investigate the effects of an adherent soft silicone anti-microbial occlusive foam silver-impregnated dressing in preventing surgical site infection (SSI) in women delivered by primary cesarean section (CS). We sought to determine if the incidence of SSIs, would be lower in patients who received a silver-impregnated dressing as compared to those who received a standard dressing, when used as part of the overall hospital protocol for reducing SSIs. Given the addition of adjunctive azithromycin antibiotic prophylaxis for those who labored or had rupture of membranes prior to undergoing a non-elective CS right at the time of initiation of the study to our institution perioperative bundle, we also elected to undertake further analyses of observational data on those with the same study inclusion criteria receiving standard dressing undergoing primary CS with subcuticular skin closure during the same time period, rather than limiting comparisons of our outcomes solely to our historical SSI rates. In order to have this comparison group, patients who declined participation in the experimental groups were selected as our non-randomized control group, given fiscal restraints precluded conducting a randomized clinical trial (RCT). Demographic, labor, delivery, intraoperative and postoperative characteristic data were collected in a de-identified fashion. Medical record review and data entry were conducted by trained research personnel. All study procedures were approved by the Investigational Review Board.

ELIGIBILITY:
Inclusion Criteria:

* Consent to undergo cesarean delivery
* Between the ages of 18 and 45
* Primary C-section
* Subcuticular skin closure
* Able to consent, fill out study documents, and complete all study procedures and follow-up visits

Exclusion Criteria:

* Patients with an allergy to silver
* Inability to obtain informed consent
* Staples
* Repeat C-section
* Vertical skin incision
* Intrapartum fever of 100F or >

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 380 (Actual)
Dates: Start 2017-07-24 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean Goodman, MD, Principal Investigator — Loyola University Chicago
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gibbs RS. Clinical risk factors for puerperal infection. Obstet Gynecol. 1980 May;55(5 Suppl):178S-184S. doi: 10.1097/00006250-198003001-00045. PMID 6990333
- [Background] Martin JA, Hamilton BE, Ventura SJ, Osterman MJ, Mathews TJ. Births: final data for 2011. Natl Vital Stat Rep. 2013 Jun 28;62(1):1-69, 72. PMID 24974591
- [Background] Owen J, Andrews WW. Wound complications after cesarean sections. Clin Obstet Gynecol. 1994 Dec;37(4):842-55. doi: 10.1097/00003081-199412000-00009. No abstract available. PMID 7842552
- [Background] National Nosocomial Infections Surveillance System. National Nosocomial Infections Surveillance (NNIS) System Report, data summary from January 1992 through June 2004, issued October 2004. Am J Infect Control. 2004 Dec;32(8):470-85. doi: 10.1016/S0196655304005425. No abstract available. PMID 15573054
- [Background] Opoien HK, Valbo A, Grinde-Andersen A, Walberg M. Post-cesarean surgical site infections according to CDC standards: rates and risk factors. A prospective cohort study. Acta Obstet Gynecol Scand. 2007;86(9):1097-102. doi: 10.1080/00016340701515225. PMID 17712651
- [Background] Vermillion ST, Lamoutte C, Soper DE, Verdeja A. Wound infection after cesarean: effect of subcutaneous tissue thickness. Obstet Gynecol. 2000 Jun;95(6 Pt 1):923-6. doi: 10.1016/s0029-7844(99)00642-0. PMID 10831993
- [Background] Culver DH, Horan TC, Gaynes RP, Martone WJ, Jarvis WR, Emori TG, Banerjee SN, Edwards JR, Tolson JS, Henderson TS, et al. Surgical wound infection rates by wound class, operative procedure, and patient risk index. National Nosocomial Infections Surveillance System. Am J Med. 1991 Sep 16;91(3B):152S-157S. doi: 10.1016/0002-9343(91)90361-z. PMID 1656747
- [Background] Yokoe DS, Christiansen CL, Johnson R, Sands KE, Livingston J, Shtatland ES, Platt R. Epidemiology of and surveillance for postpartum infections. Emerg Infect Dis. 2001 Sep-Oct;7(5):837-41. doi: 10.3201/eid0705.010511. PMID 11747696
- [Background] Declercq E, Barger M, Cabral HJ, Evans SR, Kotelchuck M, Simon C, Weiss J, Heffner LJ. Maternal outcomes associated with planned primary cesarean births compared with planned vaginal births. Obstet Gynecol. 2007 Mar;109(3):669-77. doi: 10.1097/01.AOG.0000255668.20639.40. PMID 17329519
- [Background] Cardoso Del Monte MC, Pinto Neto AM. Postdischarge surveillance following cesarean section: the incidence of surgical site infection and associated factors. Am J Infect Control. 2010 Aug;38(6):467-72. doi: 10.1016/j.ajic.2009.10.008. Epub 2010 Mar 12. PMID 20226571
- [Background] Zimlichman E, Henderson D, Tamir O, Franz C, Song P, Yamin CK, Keohane C, Denham CR, Bates DW. Health care-associated infections: a meta-analysis of costs and financial impact on the US health care system. JAMA Intern Med. 2013 Dec 9-23;173(22):2039-46. doi: 10.1001/jamainternmed.2013.9763. PMID 23999949
- [Background] Olsen MA, Butler AM, Willers DM, Gross GA, Hamilton BH, Fraser VJ. Attributable costs of surgical site infection and endometritis after low transverse cesarean delivery. Infect Control Hosp Epidemiol. 2010 Mar;31(3):276-82. doi: 10.1086/650755. PMID 20102279
- [Background] Smaill FM, Grivell RM. Antibiotic prophylaxis versus no prophylaxis for preventing infection after cesarean section. Cochrane Database Syst Rev. 2014 Oct 28;2014(10):CD007482. doi: 10.1002/14651858.CD007482.pub3. PMID 25350672
- [Background] Haas DM, Morgan S, Contreras K. Vaginal preparation with antiseptic solution before cesarean section for preventing postoperative infections. Cochrane Database Syst Rev. 2013 Jan 31;(1):CD007892. doi: 10.1002/14651858.CD007892.pub3. PMID 23440819
- [Background] Silvestry-Rodriguez N, Sicairos-Ruelas EE, Gerba CP, Bright KR. Silver as a disinfectant. Rev Environ Contam Toxicol. 2007;191:23-45. doi: 10.1007/978-0-387-69163-3_2. PMID 17708071
- [Background] Krieger BR, Davis DM, Sanchez JE, Mateka JJ, Nfonsam VN, Frattini JC, Marcet JE. The use of silver nylon in preventing surgical site infections following colon and rectal surgery. Dis Colon Rectum. 2011 Aug;54(8):1014-9. doi: 10.1097/DCR.0b013e31821c495d. PMID 21730792
- [Background] Biffi R, Fattori L, Bertani E, Radice D, Rotmensz N, Misitano P, Cenciarelli S, Chiappa A, Tadini L, Mancini M, Pesenti G, Andreoni B, Nespoli A. Surgical site infections following colorectal cancer surgery: a randomized prospective trial comparing common and advanced antimicrobial dressing containing ionic silver. World J Surg Oncol. 2012 May 23;10:94. doi: 10.1186/1477-7819-10-94. PMID 22621779
- [Background] Epstein NE. Do silver-impregnated dressings limit infections after lumbar laminectomy with instrumented fusion? Surg Neurol. 2007 Nov;68(5):483-5; discussion 485. doi: 10.1016/j.surneu.2007.05.045. PMID 17961738
- [Background] Siah CJ, Yatim J. Efficacy of a total occlusive ionic silver-containing dressing combination in decreasing risk of surgical site infection: an RCT. J Wound Care. 2011 Dec;20(12):561-8. doi: 10.12968/jowc.2011.20.12.561. PMID 22240882
- [Background] Connery SA, Downes KL, Young C. A retrospective study evaluating silver-impregnated dressings on cesarean wound healing. Adv Skin Wound Care. 2012 Sep;25(9):414-9. doi: 10.1097/01.ASW.0000419407.37323.e8. PMID 22914038
- [Background] Mangram AJ, Horan TC, Pearson ML, Silver LC, Jarvis WR. Guideline for prevention of surgical site infection, 1999. Hospital Infection Control Practices Advisory Committee. Infect Control Hosp Epidemiol. 1999 Apr;20(4):250-78; quiz 279-80. doi: 10.1086/501620. No abstract available. PMID 10219875
- [Background] Singer AJ, Arora B, Dagum A, Valentine S, Hollander JE. Development and validation of a novel scar evaluation scale. Plast Reconstr Surg. 2007 Dec;120(7):1892-1897. doi: 10.1097/01.prs.0000287275.15511.10. PMID 18090752

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment of all women admitted to labor and delivery or antepartum service to receive the silver-impregnated dressing should they deliver by primary csection
Groups:
- Silver Dressing Group: Those with primary csection and transverse incision subcuticular closure who consented to receive the silver dressing
- Standard Dressing Group: Those who had a primary csection with transverse incision subcuticular closure but who had declined to receive the silver dressing
Period: Overall Study
Arm/Group | Silver Dressing Group | Standard Dressing Group
Started | 190 | 190
Completed | 185 | 190
Not Completed | 5 | 0
Not completed — chorioamnionitis | 2 | 0
Not completed — vertical skin incision | 1 | 0
Not completed — additional dressing | 1 | 0
Not completed — never got dressing placed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Standard Dressing: Those who had a primary csection with transverse incision and subcuticular closure but who had declined to receive the silver dressing.
  Standard dressing: Telfa antimicrobial non-adherent island dressing covered with 10 sterile 4X4 gauge sponges secured wityh Tegaderm film tape. Dressing removed postop day 1 per routine.
- Total: Total of all reporting groups
Arm/Group | Silver-impregnated Antimicrobial Dressing | Standard Dressing | Total
Number analyzed (Participants) | 185 | 190 | 375
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 185 | 190 | 375
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.47 (6.34) | 29.21 (6.23) | 29.83 (6.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 185 | 190 | 375
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 41 | 56 | 97
  White | 125 | 112 | 237
  More than one race | 1 | 3 | 4
  Unknown or Not Reported | 15 | 16 | 31
Region of Enrollment [Number; unit: participants]
  United States | 185 | 190 | 375

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Wound Disruption and/or Infection
Description: Rate of wound disruption and /or infection occurring by 6 weeks was compared to a historical control rate of 10%, and to a contemporary group who received a standard dressing
Time Frame: 6 weeks postoperative
Population: 185 of original 190 who received silver dressing included in analysis. Five excluded (2 with chorioamnionitis, 1 vertical incision, 1 additional dressing applied, 1 never received silver dressing)
Measure: Count of Participants; unit: Participants
Arm/Group | Silver Dressing Group | Standard Dressing Group
Number analyzed (Participants) | 185 | 190
Participants | 5 | 9

ADVERSE EVENTS:
Time Frame: until 6 weeks postdelivery
Arm/Group | Silver Dressing Group | Standard Dressing Group
All-Cause Mortality (participants affected / at risk) | 0/185 | 0/190
Serious Adverse Events (participants affected / at risk) | 0/185 | 0/190
Other Adverse Events (participants affected / at risk) | 3/185 | 0/190
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Silver Dressing Group (N=185) | Standard Dressing Group (N=190)
pruritis (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) — itching at dressing

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-03): https://cdn.clinicaltrials.gov/large-docs/59/NCT03136159/Prot_SAP_000.pdf